CLINICAL TRIAL: NCT04216836
Title: One Week of Magnesium Supplementation Lowers IL-6, Perceived Pain and Increases Post Exercise Blood Glucose in Response to Downhill Running
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Worcester (Other)
Collaborators: Beijing Sport University (Other); Coventry University (Other)
Responsible Party: Principal Investigator, Charles Steward, Lecturer, University of Worcester
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SH17180029-R
Record Dates: First submitted 2019-09-17; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Magnesium Deficiency
Keywords: Magnesium; Supplementation; Interleukin-6; Soluble interleukin-6 receptor; Glucose; Pain; Exercise performance; Exercise recovery; Downhill running
MeSH Terms: conditions — Magnesium Deficiency; Pain | interventions — Magnesium Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High magnesium diet (SUP condition) (Experimental): Participants followed a low magnesium diet <260mg/day and consumed 500 mg/day of magnesium oxide. This was separated into 3 capsules, which were consumed at 6 hr intervals each day (8am, 2pm and 8pm). The supplementation period was 1 week.
  Interventions: Dietary Supplement: Magnesium oxide
- Low magnesium diet (CON condition) (Experimental): Participants followed a low magnesium diet <260mg/day and consumed 500 mg/day of placebo (cornflour). This was separated into 3 capsules, which were consumed at 6 hr intervals each day (8am, 2pm and 8pm). The supplementation period was 1 week.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium oxide — Magnesium capsule
  Arms: High magnesium diet (SUP condition)
Dietary Supplement: Placebo — Cornflour capsule manufactured to mimic the 166.6 mg magnesium capsule.
  Arms: Low magnesium diet (CON condition)

SUMMARY:
This study investigated the effect of magnesium supplementation on exercise performance and functional recovery in recreational endurance athletes in conjunction with measures of blood glucose, lactate, IL-6 and sIL-6R.

DETAILED DESCRIPTION:
Magnesium status can directly affect circulating glucose concentrations both during and post exercise. In addition, magnesium supplementation has been shown to reduce circulating IL-6 concentrations post exercise in humans. It is conceivable that such observations are linked through the role of IL-6 in glucose regulation, possibly in combination with sIL-6R. Together, magnesium intake may have the potential to effect exercise performance and recovery through glucose availability. This in turn may be connected to the production of IL-6 and sIL-6R which have been established to influence exercise fatigue and perception of pain (muscle soreness).

ELIGIBILITY:
Inclusion Criteria:

* Regular recreational runner, running around 3 times per week
* Capable of running 10 km in ~ 40 minutes.

Exclusion Criteria:

* Any signs or symptoms of cardiovascular issues.
* Any recent form of injury or illness.
* Currently, or in the last 3 months, have consumed multivitamin supplements
* Currently, or in the last 3 months, have consumed anti-inflammatory medications.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Downhill 10 km treadmill time trial performance | 1 day
  Maximal 10 km time trial performance on a treadmill
24 hr post exercise maximal force testing of the dominant leg on the isokinetic dynamometer | 1 day
  Maximal force produced from the dominant leg (eccentric and concentric) on an isokinetic dynamometer.

SECONDARY OUTCOMES:
Glucose | up to 2 days
  Capillary blood samples at rest, during, immediately post, 1 hr post and 24 hrs post 10 km downhill time-trial. A Biosen analyser was used to analyse glucose concentrations.
Interleukin-6 | up to 2 days
  Venous blood samples at rest, immediately post, 1hr post and 24 hrs 10 km downhill time trial. Enzyme-linked immunosorbent assays were used to analyse interleukin-6.
Soluble interleukin-6 receptor | up to 2 days
  Venous blood samples at rest, immediately post, 1hr post and 24 hrs 10 km downhill time trial. Enzyme-linked immunosorbent assays were used to analyse soluble interleukin-6.
Perceived muscle soreness | up to 4 days
  A 10cm visual analogue scale was used to assess perceived muscle soreness, the scale started at 0 (no pain) and finished at 10 (unbearable pain)
Lactate | up to 2 days
  Capillary blood samples at rest, during, immediately post, 1 hr post and 24 hrs post 10 km downhill time-trial. A Biosen analyser was used to analyse lactate concentrations.
Creatine kinase | up to 2 days
  Venous blood samples at rest, immediately post, 1hr post and 24 hrs 10 km downhill time trial. A Reflotron analyser was used to analyse creatine kinase concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Worcester, Worcester, Worcestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen HY, Cheng FC, Pan HC, Hsu JC, Wang MF. Magnesium enhances exercise performance via increasing glucose availability in the blood, muscle, and brain during exercise. PLoS One. 2014 Jan 20;9(1):e85486. doi: 10.1371/journal.pone.0085486. eCollection 2014. PMID 24465574
- [Background] Chen YJ, Chen HY, Wang MF, Hsu MH, Liang WM, Cheng FC. Effects of magnesium on exercise performance and plasma glucose and lactate concentrations in rats using a novel blood-sampling technique. Appl Physiol Nutr Metab. 2009 Dec;34(6):1040-7. doi: 10.1139/H09-105. PMID 20029512
- [Background] Cheng SM, Yang LL, Chen SH, Hsu MH, Chen IJ, Cheng FC. Magnesium sulfate enhances exercise performance and manipulates dynamic changes in peripheral glucose utilization. Eur J Appl Physiol. 2010 Jan;108(2):363-9. doi: 10.1007/s00421-009-1235-y. Epub 2009 Oct 9. PMID 19816708
- [Background] Dmitrasinovic G, Pesic V, Stanic D, Plecas-Solarovic B, Dajak M, Ignjatovic S. ACTH, Cortisol and IL-6 Levels in Athletes following Magnesium Supplementation. J Med Biochem. 2016 Nov 2;35(4):375-384. doi: 10.1515/jomb-2016-0021. eCollection 2016 Oct. PMID 28670189
- [Background] Febbraio MA, Steensberg A, Keller C, Starkie RL, Nielsen HB, Krustrup P, Ott P, Secher NH, Pedersen BK. Glucose ingestion attenuates interleukin-6 release from contracting skeletal muscle in humans. J Physiol. 2003 Jun 1;549(Pt 2):607-12. doi: 10.1113/jphysiol.2003.042374. Epub 2003 Apr 17. PMID 12702735
- [Background] Glund S, Deshmukh A, Long YC, Moller T, Koistinen HA, Caidahl K, Zierath JR, Krook A. Interleukin-6 directly increases glucose metabolism in resting human skeletal muscle. Diabetes. 2007 Jun;56(6):1630-7. doi: 10.2337/db06-1733. Epub 2007 Mar 15. PMID 17363741
- [Background] Gray SR, Ratkevicius A, Wackerhage H, Coats P, Nimmo MA. The effect of interleukin-6 and the interleukin-6 receptor on glucose transport in mouse skeletal muscle. Exp Physiol. 2009 Aug;94(8):899-905. doi: 10.1113/expphysiol.2009.048173. Epub 2009 May 29. PMID 19482899
- [Background] Robson-Ansley P, Cockburn E, Walshe I, Stevenson E, Nimmo M. The effect of exercise on plasma soluble IL-6 receptor concentration: a dichotomous response. Exerc Immunol Rev. 2010;16:56-76. PMID 20839491
- [Background] Heffernan SM, Horner K, De Vito G, Conway GE. The Role of Mineral and Trace Element Supplementation in Exercise and Athletic Performance: A Systematic Review. Nutrients. 2019 Mar 24;11(3):696. doi: 10.3390/nu11030696. PMID 30909645